CLINICAL TRIAL: NCT04027829
Title: Pharmacokinetic-pharmacodynamic Analysis for Dosing Strategy and Evaluation of Safety and Efficacy of Dexmedetomidine in Children
Brief Title: Pharmacokinetics-pharmacodynamics and Safety of Dexmedetomidine in Children
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Ministry of Food and Drug Safety, Korea (Other Government)
Responsible Party: Principal Investigator, Hee-Soo Kim, M.D., Ph.D., Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1905-188-1037
Record Dates: First submitted 2019-07-08; First posted 2019-07-22 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Intensive Care Unit; Postoperative Care
Keywords: dexmedetomidine; pediatric; sedation
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Dexmedetomidine infusion at intensive care unit
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dexmedetomidine (Experimental): Intravenous infusion of dexmedetomidine for 50 min after surgery at intensive care unit
  Interventions: Drug: Dexmedetomidine Hydrochloride

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — Intravenous infusion of dexmedetomidine at the rate of 0.5mcg/kg for 10 min, then 0.5mcg/kg/hr for 50 min.
  Other Names: Precedex

SUMMARY:
This study evaluates pharmacokinetics and pharmacodynamics of dexmedetomidine for children under sedation at intensive care unit after surgery. Patients will receive dexmedetomidine intravenously for 50 minutes after surgery as as sedation drug.

DETAILED DESCRIPTION:
Dexmedetomidine, an alpha-2 adrenergic agonist, is being effectively used for procedural sedation or sedation at intensive care unit. However, the safety and efficacy profile are not yet established for children. Although there have been some studies regrading it, still there is no public guideline, therefore making it difficult to use dexmedetomidine in children.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients planned to undergo mechanical ventilation at intensive care unit after surgery
* Pediatric patients planned to be extubated within 4 hours after surgery for neurological examination
* Patients whose parent of legal guardian agreed to enroll in the study after having enough time to review the complete explanation about the study.

Exclusion Criteria:

* History of hypersensitivity to any drugs including dexmedetomidine.
* Underlying cardiovascular/circulatory disease
* Underlying liver / kidney disease
* Patients under hemodialysis
* Obesity of BMI > 35
* Patients planned to receive patient-controlled analgesia including opioids
* Patients whose parent or legal guardian declined to enroll in the study
* Other conditions deemed unsuitable for the study

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2019-08-14 (Actual); Primary Completion 2019-11-14 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of dexmedetomidine | From start of dexmedetomidine infusion to 480 minutes after end of dexmedetomidine infusion
  Plasma concentration of dexmedetomidine before infusion, 10/30/60 minutes after initiation of infusion, 15/30/60/120/240/480 minutes after end of infusion
Bispectral index | From start of dexmedetomidine infusion to 480 minutes after end of dexmedetomidine infusion
  Bispectral index based on electroencephalogram during patient's stay at intensive care unit (0-100, lower score implies deeper sedation)
University of Michigan Sedation Scale | From start of dexmedetomidine infusion to 480 minutes after end of dexmedetomidine infusion
  University of Michigan Sedation Scale based on observer's inspection during patient's stay at intensive care unit (0-4, higher score implies deeper sedation)

SECONDARY OUTCOMES:
Incidence of arrhythmia | From start of dexmedetomidine infusion to 24 hours after end of dexmedetomidine infusion
  Presence of any kind of arrhythmia from electrocardiogram following dexmedetomidine infusion
Non-invasive blood pressure | From start of dexmedetomidine infusion to 24 hours after end of dexmedetomidine infusion
  Non-invasive blood pressure in units of mmHg, to examine whether hypertension (increase in blood pressure more than 20% of baseline) or hypotension (decrease in blood pressure more than 20% of baseline) occurs
Incidence of desaturation | From start of dexmedetomidine infusion to 24 hours after end of dexmedetomidine infusion
  Presence of desaturation (pulse oximetry of lower than 94%) following dexmedetomidine infusion
Respiratory rate | From start of dexmedetomidine infusion to 24 hours after end of dexmedetomidine infusion
  Respiratory rate in units of /min, to examine whether respiratory depression or apnea occurs
Incidence of nausea | From start of dexmedetomidine infusion to 24 hours after end of dexmedetomidine infusion
  Incidence of nausea following dexmedetomidine infusion
Incidence of vomiting | From start of dexmedetomidine infusion to 24 hours after end of dexmedetomidine infusion
  Incidence of vomiting following dexmedetomidine infusion

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, M.D., Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongro Gu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tobias JD. Dexmedetomidine: applications in pediatric critical care and pediatric anesthesiology. Pediatr Crit Care Med. 2007 Mar;8(2):115-31. doi: 10.1097/01.PCC.0000257100.31779.41. PMID 17273114
- [Background] Su F, Hammer GB. Dexmedetomidine: pediatric pharmacology, clinical uses and safety. Expert Opin Drug Saf. 2011 Jan;10(1):55-66. doi: 10.1517/14740338.2010.512609. Epub 2010 Aug 18. PMID 20718689
- [Background] Reiter PD, Pietras M, Dobyns EL. Prolonged dexmedetomidine infusions in critically ill infants and children. Indian Pediatr. 2009 Sep;46(9):767-73. Epub 2009 Apr 1. PMID 19430081
- [Background] Banasch HL, Dersch-Mills DA, Boulter LL, Gilfoyle E. Dexmedetomidine Use in a Pediatric Intensive Care Unit: A Retrospective Cohort Study. Ann Pharmacother. 2018 Feb;52(2):133-139. doi: 10.1177/1060028017734560. Epub 2017 Sep 27. PMID 28952341
- [Background] Sulton C, McCracken C, Simon HK, Hebbar K, Reynolds J, Cravero J, Mallory M, Kamat P. Pediatric Procedural Sedation Using Dexmedetomidine: A Report From the Pediatric Sedation Research Consortium. Hosp Pediatr. 2016 Sep;6(9):536-44. doi: 10.1542/hpeds.2015-0280. Epub 2016 Aug 11. PMID 27516413
- [Background] Plambech MZ, Afshari A. Dexmedetomidine in the pediatric population: a review. Minerva Anestesiol. 2015 Mar;81(3):320-32. Epub 2014 May 14. PMID 24824958
- [Background] Kim HS, Byon HJ, Kim JE, Park YH, Lee JH, Kim JT. Appropriate dose of dexmedetomidine for the prevention of emergence agitation after desflurane anesthesia for tonsillectomy or adenoidectomy in children: up and down sequential allocation. BMC Anesthesiol. 2015 May 27;15:79. doi: 10.1186/s12871-015-0059-z. PMID 26012345
- [Background] Mahmoud M, Mason KP. Dexmedetomidine: review, update, and future considerations of paediatric perioperative and periprocedural applications and limitations. Br J Anaesth. 2015 Aug;115(2):171-82. doi: 10.1093/bja/aev226. PMID 26170346
- [Background] Tobias JD, Berkenbosch JW. Sedation during mechanical ventilation in infants and children: dexmedetomidine versus midazolam. South Med J. 2004 May;97(5):451-5. doi: 10.1097/00007611-200405000-00007. PMID 15180019
- [Background] Chrysostomou C, Sanchez De Toledo J, Avolio T, Motoa MV, Berry D, Morell VO, Orr R, Munoz R. Dexmedetomidine use in a pediatric cardiac intensive care unit: can we use it in infants after cardiac surgery? Pediatr Crit Care Med. 2009 Nov;10(6):654-60. doi: 10.1097/PCC.0b013e3181a00b7a. PMID 19295456
- [Background] Walker J, Maccallum M, Fischer C, Kopcha R, Saylors R, McCall J. Sedation using dexmedetomidine in pediatric burn patients. J Burn Care Res. 2006 Mar-Apr;27(2):206-10. doi: 10.1097/01.BCR.0000200910.76019.CF. PMID 16566567
- [Background] Koroglu A, Demirbilek S, Teksan H, Sagir O, But AK, Ersoy MO. Sedative, haemodynamic and respiratory effects of dexmedetomidine in children undergoing magnetic resonance imaging examination: preliminary results. Br J Anaesth. 2005 Jun;94(6):821-4. doi: 10.1093/bja/aei119. Epub 2005 Mar 11. PMID 15764627
- [Background] Berkenbosch JW, Wankum PC, Tobias JD. Prospective evaluation of dexmedetomidine for noninvasive procedural sedation in children. Pediatr Crit Care Med. 2005 Jul;6(4):435-9; quiz 440. doi: 10.1097/01.PCC.0000163680.50087.93. PMID 15982430
- [Background] Chrysostomou C, Schulman SR, Herrera Castellanos M, Cofer BE, Mitra S, da Rocha MG, Wisemandle WA, Gramlich L. A phase II/III, multicenter, safety, efficacy, and pharmacokinetic study of dexmedetomidine in preterm and term neonates. J Pediatr. 2014 Feb;164(2):276-82.e1-3. doi: 10.1016/j.jpeds.2013.10.002. Epub 2013 Nov 14. PMID 24238862
- [Background] Diaz SM, Rodarte A, Foley J, Capparelli EV. Pharmacokinetics of dexmedetomidine in postsurgical pediatric intensive care unit patients: preliminary study. Pediatr Crit Care Med. 2007 Sep;8(5):419-24. doi: 10.1097/01.PCC.0000282046.66773.39. PMID 17693909